CLINICAL TRIAL: NCT07049601
Title: Effect of Tight Glycemic Control on Microvascular Complications in Type 2 Diabetes Mellitus: A Randomized Controlled Trial in an Egyptian Cohort
Brief Title: THE Effect of Tight Glycemic Control on Microvascular Complications in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Moustafa Shaheen, Assistant Lecturer of Internal Medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FMASU MD 119/2022
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus
Keywords: tight glycemic control
MeSH Terms: conditions — Diabetes Mellitus | interventions — Convulsive Therapy; Hypoglycemic Agents; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tight glycemic control (Active Comparator): Patients received treatment through insulin therapy, oral hypoglycemics and lifestyle and nutrition education to achieve tight glycemic control with HbA1c less than 7%
  Interventions: Other: Insulin Therapy; Other: Antidiabetic therapy, lifestyle modification
- Less tight glycemic control (Active Comparator): Patients received treatment through insulin therapy, oral hypoglycemics and lifestyle and nutrition education to achieve tight glycemic control with HbA1c less than 7.5
  Interventions: Other: Insulin Therapy; Other: Antidiabetic therapy, lifestyle modification

INTERVENTIONS:
Other: Insulin Therapy — The effect of this intervention on HbA1c leading to either tight glycemic control HbA1c less than 7% or less tight glycemic control HbA1c less than 7.5%
  Other Names: oral antidiabetics; lifestyle and nutrition education
Other: Antidiabetic therapy, lifestyle modification — Individualized adjustments in antidiabetic therapy, lifestyle modification, and monthly clinical follow-up.

SUMMARY:
The goal of this clinical trial is to learn the impact of tight versus less tight glycemic control on microvascular complications among Egyptian adults with uncontrolled T2DM. The main question it aims to answer is:

Does tight glycemic control improve or worsens microvascular complications of diabetes compared to less tight glycemic control?

Participants will:

* Be divided to two groups according to their HbA1c group A tight glycemic control and less tight glycemic control.
* Be followed for 6 months with clinical, laboratory, and fundoscopic evaluations performed at baseline and endpoint.

DETAILED DESCRIPTION:
Background: Tight glycemic control is widely promoted in the management of type 2 diabetes mellitus (T2DM) to reduce microvascular complications, yet the extent and speed of HbA1c reduction may paradoxically exacerbate certain outcomes.

Objective: To assess the impact of tight versus less tight glycemic control on microvascular complications among Egyptian adults with uncontrolled T2DM.

Methods: In this randomized controlled trial, 80 patients with poorly controlled T2DM (HbA1c >7.5%) were randomized into two groups: Group A (tight control, HbA1c <7.0%) and Group B (less tight control, HbA1c <7.5%). Participants were followed for 6 months with clinical, laboratory, and fundoscopic evaluations performed at baseline and endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Age 18-60years old.
* Patients diagnosed with Diabetes Mellitus (Type 2) according to American Diabetes Association (ADA) guidelines.
* Patients willing to participate after signing a written consent to be enrolled in the study after being explained to them in an interview.
* Diabetic patients with mild and moderate non proliferative diabetic retinopathy

Exclusion Criteria:

* Patients with age above 60 or below 18 years old.
* Patients with severe non proliferative diabetic retinopathy up to advanced proliferative diabetic retinopathy.
* Patients diagnosed with type 1 DM.
* Patients with malignant tumours.
* Patients with end stage renal disease and end stage liver disease.
* Patients with history of myocardial infarction.
* Patients with recurrent attacks of hypoglycemia and hypoglycemia unawareness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Effect of Tight Glycemic Control on Microvascular Complications (Retinopathy, neuropathy and Nephropathy) in Type 2 Diabetes Mellitus in 80 patients divided into two groups according to their HbA1c | 18 months
  80 patients with poorly controlled T2DM (HbA1c >7.5%) were randomized into two groups according to their HbA1c: Group A (tight control, HbA1c <7.0%) and Group B (less tight control, HbA1c <7.5%). Participants were followed for 6 months with clinical, laboratory and fundoscopic evaluations performed at baseline and endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Professor of internal medicine and endocrinology, Study Director — Ain Shams University; Assistant Professor of internal medicine and endocrinology, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT07049601/Prot_000.pdf